CLINICAL TRIAL: NCT06877806
Title: Effects of Core Exercise on Posture and Trunk Endurance Parameters in Sedentary Males: A Randomized Controlled Trial
Brief Title: Effects of Core Exercise on Posture and Trunk Endurance in Sedentary Males
Acronym: Coremale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Dragan Marinkovic, Principal investigator, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/2018
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Posture; Trunk Muscle Endurance
Keywords: Core exercise; Sedentary males; Posture; Trunk endurance; Neuromuscular improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Core Exercise (Experimental): Core exercise and trunk endurance intervention
  Interventions: Other: Core exercise
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Core exercise — The experimental treatment had a total of 18 introductory courses lasting 30 minutes each. The treatment included exercises to increase the mobility and strength of the neck, shoulders, pelvis and hips, and anti-flexion, anti-extension and rotation exercises were used to stabilize the spine. McGill curl-up was performed during each treatment for all 6 weeks. In the first two weeks, the subjects did general and introductory exercises (all positioned planks, plank walking, forearm cranes, plank pad forearms, etc.). Week 3 and 4 with additional movements and rotations (alternating hand and foot board holding, superman posture, faceplate switches, etc.). During the fifth and sixth weeks, the exercises were performed on unstable surfaces (one-handed board, ball stirring pot, feet raised sideboard, etc.). The intensity of those training courses was individual, but each one started at submaximal.
  Arms: Core Exercise

SUMMARY:
Increased sedentary lifestyles due to modern technological advancements have negatively impacted posture and trunk stability. Proper posture relies on balanced dorsal and ventral muscles, trunk stabilization, and joint flexibility. Deviations in these factors may lead to postural abnormalities and, over time, structural deformities. Early detection and intervention through corrective exercises can mitigate these issues. Various measurement techniques, including 2D and 3D scanning, allow for objective posture assessment. Core stabilization exercises have been shown to influence spinal alignment and muscle endurance, improving postural control. However, limited research focuses on young adult males. This study aimed to evaluate the effects of an 8-week core exercise program on posture and trunk endurance in sedentary university students.

A randomized controlled trial was conducted on male university students at the University of Novi Sad, Serbia. Participants were recruited through an open call, and those with prior musculoskeletal, neurological, or metabolic conditions were excluded. The final sample included 138 participants divided into an experimental group (EG) and a control group (CG). The EG followed an 8-week core stabilization program, while the CG did not receive any intervention.

Postural assessments were conducted using CONTEMPLAS TEMPLO software with 2D and 3D analysis protocols. Measurements included the Fröner Posture Index (PI) and the Kyphosis-Inclination-Lordosis (KIL) scheme, evaluating thoracic kyphosis, cervico-lumbar, and lumbar-gluteal angles. Trunk endurance was assessed through the Sorensen Back Extensor Test (BET), the Abdominal Flexor Endurance Test (FET), and the Double Leg Lowering Test (DLL). The intervention program consisted of progressive core stabilization exercises, increasing in difficulty from basic planks to exercises on unstable surfaces.

The experimental group underwent structured core training three times a week for eight weeks. The program included exercises to enhance mobility and strengthen the neck, shoulders, pelvis, and hips, with a focus on stabilizing the spine through anti-flexion, anti-extension, and anti-rotation movements. Exercises progressed from static planks to dynamic and unstable surface training. The control group did not participate in any structured physical activity.

DETAILED DESCRIPTION:
At the beginning of the 21st century, technological and social changes have significantly impacted human health and development. Increased reliance on technology has contributed to a sedentary lifestyle, leading to reduced physical activity and associated health issues. One major concern is the effect of prolonged sitting on posture and trunk stability. Proper posture is essential for maintaining musculoskeletal health and functional movement. It depends on the balance between dorsal and ventral muscles, the strength of trunk stabilizers, and the flexibility of joints.

Misalignments in body posture, especially in the sagittal plane, can lead to postural abnormalities. If left untreated, these abnormalities may develop into structural deformities. The biomechanics of the spine are particularly sensitive to prolonged external forces, which can result in muscular imbalances and impaired postural reflexes. Addressing these issues through early intervention and corrective exercises can help restore proper alignment and reduce the risk of developing chronic conditions.

Traditional postural assessments often rely on visual inspection, which lacks scientific precision. Recent advancements in technology, such as 2D and 3D scanning techniques, allow for more objective posture evaluation. The CONTEMPLAS TEMPLO software is one such tool that provides detailed postural analysis based on reference points, angles, and postural indices. Using such technologies, researchers can quantitatively assess changes in posture before and after intervention programs.

Several studies have demonstrated the benefits of core stabilization exercises in improving postural control and trunk endurance. These exercises have been shown to correct thoracic and lumbar curvatures, enhance muscular balance, and improve movement patterns. However, most posture-related studies focus on children and adolescents. There is limited research on postural interventions in young adult males. The present study aims to investigate the effects of an 8-week core exercise program on posture and trunk endurance in sedentary university students.

The study recruited male university students from the University of Novi Sad, Serbia. Participants were selected through an open application process, with an initial sample of 250 individuals. After an initial screening, 230 participants met the inclusion criteria. The selection process was designed to ensure a homogeneous sample by excluding individuals with prior musculoskeletal, neurological, or metabolic conditions that could affect balance and posture.

After randomization, 230 participants were divided into two groups:

Measurements Anthropometric Measurements Height: Measured using Martin's anthropometry Weight: Measured using a digital scale BMI: Calculated based on height and weight Postural Assessment Postural disorders were evaluated using the CONTEMPLAS TEMPLO photometric system, which analyzes body alignment based on 2D and 3D protocols.

2D Analysis Fröner Posture Index (PI): Calculated based on spinal curvatures, including thoracic kyphosis and lumbar lordosis. PI values range from 0.8 to 1.7, with optimal posture between 1.0 and 1.2.

Kyphosis-Inclination-Lordosis (KIL) Scheme: Evaluates:

Thoracic Kyphosis Index (TKI) Cervico-Lumbar Lead Angle (CCL) Lumbar-Gluteal Lead Angle (LGL) The KIL scheme helps assess postural asymmetry and spinal curvatures.

3D Analysis

The 3D spine analysis protocol provides a comprehensive assessment of the sagittal and frontal posture, including:

Shoulder and pelvis alignment Spinal curvature relative to the vertical reference line

Trunk Muscle Endurance Tests Sorensen Back Extensor Test (BET): Measures back extensor endurance in a prone position. Participants attempt to maintain a horizontal position for as long as possible.

Abdominal Flexor Endurance Test (FET): Measures abdominal endurance with participants sitting at a 50-degree incline and maintaining the position.

Double Leg Lowering Test (DLL): Assesses core stability by measuring the angle at which participants can control pelvic movement during leg lowering.

Intervention Protocol

Control Group (CG) The control group received no intervention and continued their regular daily activities.

Experimental Group (EG)

The experimental group participated in an 8-week core stabilization program, conducted three times per week. Each session lasted 30 minutes and consisted of:

Weeks 1-2:

Basic stabilization exercises (planks, forearm support, quadruped positioning) Core activation drills (McGill curl-up, plank walking)

Weeks 3-4:

Additional movement patterns (superman holds, alternating hand and foot raises) Rotation-based stabilization (faceplate switches)

Weeks 5-6:

Introduction of unstable surfaces (stability ball, balance boards) Unilateral exercises (single-leg planks, single-arm support)

Weeks 7-8:

Advanced core exercises (stirring the pot, one-arm side planks) Increased resistance and endurance-based progressions The intensity of the program was gradually increased based on participants' progress.

ELIGIBILITY:
Inclusion Criteria:

* no injuries within the past six months,
* no other medical conditions, including COVID-19,
* no scheduled physical activity in the previous three months,
* we considered the experimental programs valid if participants completed at least 80% of all training sessions.

Exclusion Criteria:

* had a history of neurological or musculoskeletal disorders,
* had clinical conditions that could affect balance, such as motor disorders, diabetes, heart disease, stroke, vision problems, thyroid issues, or issues with nerves or blood vessels.

Ages: 19 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
3D Cervical | 6 weeks
  Postural disorders were evaluated using the CONTEMPLAS TEMPLO photometric system, which analyses body alignment-based 3D protocols. Markers were set on anatomical landmark: CV7 - Cervical Vertebrae 7 and SACR - Sacrum and system calculate distance cervical spine - sacrum. Distance indicates the cervical spine regarding the vertical line projection of the sacrum (the bone at the bottom of the spine) in the sagittal plane. Values are presented in centimeters (cm).
3D Thoracic | 6 weeks
  Postural disorders were evaluated using the CONTEMPLAS TEMPLO photometric system, which analyses body alignment-based 3D protocols. Markers were set on anatomical landmark: MAI - Midpoint Between the Inferior Angles of Most Caudal Points of the Two Scapula and SACR - Sacrum and system calculate distance thoracic spine - sacrum. Distance indicates the thoracic spine regarding the vertical line projection of the sacrum (the bone at the bottom of the spine) in the sagittal plane. Values are presented in centimeters (cm).
3D Lumbar | 6 weeks
  Postural disorders were evaluated using the CONTEMPLAS TEMPLO photometric system, which analyses body alignment-based 3D protocols. Markers were set on anatomical landmark: LV1 - Lumbar Level Vertebrae 1 and SACR - Sacrum and system calculate distance Lumbar spine - sacrum. Distance indicates the lumbar (lower) spine regarding the vertical line projection of the sacrum (the bone at the bottom of the spine) in the sagittal plane. Values are presented in centimeters (cm).
Thoracic kyphosis Index (TKI) | 6 weeks
  Postural disorders were evaluated using the CONTEMPLAS TEMPLO photometric system, which analyses body alignment-based 2D protocols. Markers were set on anatomical landmark: C - Cervical Vertebrae 7; D - Midpoint Between the Inferior Angles of Most Caudal Points of the Two Scapula; L - Lumbar Level Vertebrae 1; G - Maximal present point of gluteus; D1 - Vertical projection that connect line from Cervical point to Lumbar point.
  TKI=(D*D1)*25/ distance from C to L; Values: Optimal 2,3 to 3,0; Acceptable 3,1 to 4,0; Marginal 4,1 to 4,4; Suspicious 4,5 to 5,0; Conspicuous more than 5,0.
Cervical-lumbar lead angle (CLL) | 6 weeks
  Postural disorders were evaluated using the CONTEMPLAS TEMPLO photometric system, which analyses body alignment-based 2D protocols. Markers were set on anatomical landmark: C - Cervical Vertebrae 7; D - Midpoint Between the Inferior Angles of Most Caudal Points of the Two Scapula; L - Lumbar Level Vertebrae 1; G - Maximal present point of gluteus; D1 - Vertical projection that connect line from Cervical point to Lumbar point. CLL angle was measured at point L. It presents the angle between the perpendicular and the connection line of point L and C. It describes the sagittal inclination of the spine. Values: Optimal --2 to 1; Acceptable -2 to -6; Marginal -7 to -8; Suspicious -9 to -10,5; Conspicuous less than -10,5.
Lumbar-gluteal lead angle (LGL) | 6 weeks
  Postural disorders were evaluated using the CONTEMPLAS TEMPLO photometric system, which analyses body alignment-based 2D protocols. Markers were set on anatomical landmark: C - Cervical Vertebrae 7; D - Midpoint Between the Inferior Angles of Most Caudal Points of the Two Scapula; L - Lumbar Level Vertebrae 1; G - Maximal present point of gluteus; D1 - Vertical projection that connect line from Cervical point to Lumbar point. Was measured at point G. The angle between the connection line of Point L to G and the perpendicular to point G. It is the measured values for the lordosis. Values: Optimal -10 to -23; Acceptable -24 to -28; Marginal -29 to -31; Suspicious -32 to -35; Conspicuous less than -36.
Sorensen Back Extensor Test (BET) | 6 weeks
  The Sorensen Back Extensor Test (BET) assesses back extensor endurance. The subject lies prone on a table with the iliac crest aligned to the edge. The lower body is secured with straps while the upper body extends unsupported over the edge. With arms crossed over the chest, the subject maintains a horizontal position as long as possible. The test ends when the subject can no longer hold the position due to fatigue or pain. The time (in seconds) is recorded, with longer durations indicating better endurance.
Abdominal Flexor Endurance Test (FET) | 6 weeks
  The Abdominal Flexor Endurance Test (FET) assesses core endurance. The subject sits with knees bent at 90 degrees, feet flat, and arms crossed over the chest. The upper body leans back to a 60-degree angle from the floor. Once support is removed, the subject must hold this position without moving or arching. The test ends when the subject can no longer maintain the posture. Time (in seconds) is recorded, with longer durations indicating better abdominal endurance.
Double Leg Lowering Test (DLL) | 6 weeks
  The Double Leg Lowering Test (DLL) assesses lower abdominal and core strength. The subject lies supine with arms at the sides and legs raised to a 90-degree hip flexion. While keeping the lower back in contact with the floor, the subject slowly lowers both legs until they can no longer maintain pelvic control or lumbar stability. The angle at which the back arches or control is lost is recorded. A lower angle indicates better core strength, while early loss of control suggests weakness.

SECONDARY OUTCOMES:
Age | 6 weeks
  The participant's date of birth is collected in order to calculate his age in years.
Weight | 6 weeks
  The weight of the participants is analyzed in kilograms.
Height | 6 weeks
  The height of the subject is determined in meters.
Body Mass Index (BMI) | 6 weeks
  The participant's BMI is calculated from his height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Marinkovic, Msc, Principal Investigator — University of Novi Sad, Faculty of Sport and Physical Education
Locations (1):
- University of Novi Sad, Faculty of Sport and Physical Education, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: No